CLINICAL TRIAL: NCT01495637
Title: GM-CSF for Immunomodulation Following Trauma (GIFT) Study
Acronym: GIFT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mark Hall (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Mark Hall, Professor of Pediatrics, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIFT Study; R01GM094203 (NIH); UG1HD083170 (NIH)
Record Dates: First submitted 2011-12-13; First posted 2011-12-20 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Critical Injury (Trauma) in Children
Keywords: pediatric; trauma; critical; GM-CSF; immune
MeSH Terms: conditions — Wounds and Injuries | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GM-CSF (Experimental): GM-CSF is given in one of four treatment regimens (three days at a dose of 30, 62, or 125 mcg/m2/day, or extended dosing at 125 mcg/m2 through post-trauma day 6) to critically injured children who demonstrate severe reduction in innate immune function on post-trauma day 1, 2, or 3.
  Interventions: Drug: GM-CSF

INTERVENTIONS:
Drug: GM-CSF — GM-CSF is to be administered IV at one of four possible dosing regimens (three days at a dose of 30, 62, or 125 mcg/m2 per day, or an extended dosing regimen of 125 mcg/m2/day through post-trauma 6) if severe innate immune suppression is identified on post-trauma days 1, 2, or 3.
  Other Names: sargramostim; leukine

SUMMARY:
The GIFT study is a prospective, multi-center, interventional trial using the drug GM-CSF for the reversal of innate immune suppression in critically injured children. The study will be conducted in two phases, a dose-finding phase then an efficacy phase. The dose-finding phase is the current active phase of the study. The central hypothesis of the study is that immunomodulation with GM-CSF will result in reduction in the risk of nosocomial infection after critical injury in high-risk children through safe, rapid, and sustained improvement in innate immune function.

DETAILED DESCRIPTION:
The current phase of the study is an open-label dose-finding phase in which critically injured children undergo prospective, serial immune function testing in the first few days after injury. If a subject's immune function (as measured by whole blood ex vivo LPS-induced TNF-alpha production capacity) is below a critical threshold, the subject will receive GM-CSF at a dose of 30, 62, or 125 mcg/m2 per day for three days. Enrollment is stratified by pubertal status (Tanner 1 or Tanner > 1) and by presence or absence of severe traumatic brain injury (TBI). Dose-finding is being conducted independently in each of these strata. The outcome variable for the dose-finding phase of the GIFT study is restoration of TNF-alpha production capacity and monocyte HLA-DR expression by the end of treatment, persisting to post-trauma day 7. A subsequent randomized, placebo-controlled trial with nosocomial infection as the primary outcome variable is planned once dose-finding is complete. This study is being conducted by the NICHD's Collaborative Pediatric Critical Care Research Network (CPCCRN) with Nationwide Children's Hospital as the primary site. The study design information currently displayed on this site refers to the dose-finding phase of the project.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the PICU at a GIFT study site with a primary diagnosis of blunt or penetrating trauma that occurred within the last 72 hours.
* Age 1 - 17 years
* Provisional Injury Severity Score (ISS) > 10
* Presence of an endotracheal tube at the time of enrollment

Exclusion Criteria:

* DNR status or care team/family is considering plans for withdrawal of life-sustaining therapies.
* Strong suspicion of injuries related to child abuse, in the opinion of the treating physician
* Persistence (after treatment) of any of the following in the PICU before enrollment: Fixed, dilated pupils; Glasgow Coma Scale score of 3 (in the absence of neuromuscular blocking drugs); or presence of a new, severe neurologic injury at the time of enrollment which, in the opinion of the treating physician, is highly likely to lead to a diagnosis of brain death
* Cardiopulmonary arrest requiring CPR documented by EMS or hospital personnel prior to subject identification
* Burn injury of any kind (scald, fire, chemical)
* Patients receiving acute or chronic immunosuppressive therapy (e.g., systemic corticosteroids, calcineurin inhibitors, mycophenolate, azathioprine) at the time of injury
* Patients with severe leukopenia (white blood cell count < 1000 cells/mm3) at the time of injury as the result of myeloablative chemotherapy or radiation
* Pregnancy
* Autoimmune thrombocytopenia, myelodysplastic syndromes with > 20% marrow blast cells, or known allergy/hypersensitivity to GM-CSF
* Previously enrolled in the GIFT study

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2022-02 (Actual); Study Completion 2023-02 (Actual)

PRIMARY OUTCOMES:
Immune function | 7-days post-trauma
  To identify the lowest immunostimulatory yet tolerable dose of GM-CSF that produces lasting improvement in innate immune function in treated children.

SECONDARY OUTCOMES:
Nosocomial infection | 28-days post-trauma
  The development of hospital-acquired infection through post-trauma day 28

CONTACTS AND LOCATIONS:
Overall Officials: Mark W Hall, MD, Principal Investigator — Nationwide Children's Hospital
Locations (8):
- United States (8):
  - Children's Hospital of Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Hospital of Michigan, Detroit, Michigan
  - Washington University / St. Louis Children's Hospital, St Louis, Missouri
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
A public use data set will be made available on the website of the NICHD's Collaborative Pediatric Critical Care Research Network.
Supporting Information: Study Protocol, CSR
Time Frame: Within one year of study completion.
Access Criteria: Access is through web request on the CPCCRN website